CLINICAL TRIAL: NCT02701257
Title: The iLet Introduction Study: A Feasibility Study of the iLet, a Fully Integrated Bihormonal Bionic Pancreas
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated prior to completing the planned cohorts and analysis because of problems with the infusion set resulting in inadequate insulin delivery
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015P002773
Record Dates: First submitted 2016-02-29; First posted 2016-03-08 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus Type 1
Keywords: Bionic Pancreas; Insulin; Glucagon; Continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- iPhone bionic pancreas - Lilly glucagon (Active Comparator): iPhone based bionic pancreas using insulin lispro and Lilly glucagon. These visits will be conducted separately from the infusion set sub-study visits.
  Interventions: Device: iPhone bionic pancreas; Drug: Lilly glucagon
- iLet bionic pancreas - Lilly glucagon (Experimental): iLet Bionic Pancreas using using insulin lispro and Lilly glucagon. These visits will be conducted separately from the infusion set sub-study visits.
  Interventions: Device: iLet bionic pancreas; Drug: Lilly glucagon
- iLet bionic pancreas - Xerisol glucagon (Experimental): iLet Bionic Pancreas using using insulin lispro and Xeris Xerisol glucagon. These visits will be conducted separately from the infusion set sub-study visits.
  Interventions: Device: iLet bionic pancreas; Drug: Xeris Xerisol glucagon
- iLet infusion set (Experimental): The infusion set sub-study will be testing just the experimental iLet infusion set in a crossover with the contact detach infusion set. These visits will be conducted separately from the iPhone and iLet bionic pancreas visits.
  Interventions: Device: iLet infusion set
- Contact Detach infusion set (Active Comparator): The infusion set sub-study will be testing just the experimental iLet infusion set in a crossover with the contact detach infusion set. These visits will be conducted separately from the iPhone and iLet bionic pancreas visits.
  Interventions: Device: Contact Detach infusion set

INTERVENTIONS:
Device: iPhone bionic pancreas — An experimental device composed of three parts: a continuous glucose monitor, control algorithms running on an iPhone, and drug delivery using Tandem insulin pumps
  Arms: iPhone bionic pancreas - Lilly glucagon
Device: iLet bionic pancreas — An experimental device that combines the functions of the iPhone-based bionic pancreas into one device.
  Arms: iLet bionic pancreas - Lilly glucagon; iLet bionic pancreas - Xerisol glucagon
Drug: Xeris Xerisol glucagon — A stabilized formulation of human glucagon in a solvent based primarily composed of dimethyl sulfoxide (DMSO) that has prolonged stability and can be used for multiple days in a pump
  Other Names: Xeris glucagon
  Arms: iLet bionic pancreas - Xerisol glucagon
Drug: Lilly glucagon — An aqueous formulation of human glucagon with limited stability that must be changed daily
  Other Names: glucagon
  Arms: iLet bionic pancreas - Lilly glucagon; iPhone bionic pancreas - Lilly glucagon
Device: iLet infusion set — The infusion set sub-study will be studying the experimental iLet infusion set in a cross-over with the Contact Detach infusion set. These visits will be conducted separately from the iPhone and iLet BP visits.
  Arms: iLet infusion set
Device: Contact Detach infusion set — The infusion set sub-study will be studying the experimental iLet infusion set in a cross-over with the Contact Detach infusion set. These visits will be conducted separately from the iPhone and iLet BP visits.
  Arms: Contact Detach infusion set

SUMMARY:
This study will compare two different models of a wearable bionic pancreas device (the iPhone-based bionic pancreas vs. the iLet bionic pancreas) in adult participant with type 1 diabetes. Both bionic pancreas devices measure glucose levels every five minutes and then give insulin and/or glucagon automatically to regulate the blood glucose (BG).

DETAILED DESCRIPTION:
The iPhone bionic pancreas has been used in earlier studies, during which volunteers used the system for up to 11 days at a time while living their normal lives at home and work. The iLet bionic pancreas has never been tested in humans. In this new study, volunteers will participate in a training visit to learn how both devices work. They will then use the iPhone-based BP for 1 day and the iLet BP for 1 day in random order using Lilly glucagon. They will then use the iLet BP for one additional day using Xeris Xerisol glucagon (a stable formulation of human glucagon).

A custom infusion set is required for this bihormonal system, to prevent future consumers from being able to accidentally swap their insulin and glucagon reservoirs and infusion sets, which could be potentially fatal. Previous experiments have demonstrated flaws in the infusion set design, requiring human experiments to be suspended and modifications to the infusion set be made. We believe the current infusion set has addressed these flaws by incorporating an anti-coring heel and a tri-beveled needle, and the infusion set sub-study is designed to isolate and study the infusion set function before further experiments using the iLet BP are conducted.

ELIGIBILITY:
Inclusion Criteria:

iPhone and iLet BP experiments

* Age ≥ 18 years and have had clinical type 1 diabetes for at least one year
* Diabetes managed using an insulin pump for ≥ 6 months
* Prescription medication regimen stable for > 1 month (except for medications that will not affect the safety of the study and are not expected to affect any outcome of the study, in the judgment of the principal investigator)

iLet Infusion Set Sub-Study

* Age ≥ 18 years and have had clinical type 1 diabetes for at least one year
* Diabetes managed using an insulin pump for ≥ 6 months

Exclusion Criteria:

iPhone and iLet BP experiments

* Unable to provide informed consent (e.g. impaired cognition or judgment)
* Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the bionic pancreas, impaired memory, unable to speak and read English)
* Current participation in another diabetes-related clinical trial that, in the judgment of the principal investigator, will compromise the results of this study or the safety of the subject
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception
* Current alcohol abuse (intake averaging > 3 drinks daily in last 30 days), use of marijuana within 1 month of enrollment, or other substance abuse (use within the last 6 months of controlled substances other than marijuana without a prescription)
* Unwilling or unable to refrain on the study days from:acetaminophen in any form, use of marijuana, use of drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study (use of beta blockers will be allowed as long as the dose is stable and the subject does not meet the criteria for hypoglycemia unawareness while taking that stable dose, but use of benzodiazepines or narcotics, even if by prescription, may be excluded according to the judgment of the principal investigator)
* History of liver disease that is expected to interfere with the anti-hypoglycemia action of glucagon (e.g. liver failure or cirrhosis). Other liver disease (i.e. active hepatitis, steatosis, active biliary disease, any tumor of the liver, hemochromatosis, glycogen storage disease) may exclude the subject if it causes significant compromise to liver function or may do so in an unpredictable fashion.
* Renal failure on dialysis
* Personal history of cystic fibrosis, pancreatitis, pancreatic tumor, or any other pancreatic disease besides type 1 diabetes
* Any known history of coronary artery disease including, but not limited to, history of myocardial infarction, stress test showing ischemia, history of angina, or history of intervention such as coronary artery bypass grafting, percutaneous coronary intervention, or enzymatic lysis of a presumed coronary occlusion)
* Congestive heart failure (established history of CHF, lower extremity edema, paroxysmal nocturnal dyspnea, or orthopnea)
* History of TIA or stroke
* Seizure disorder, history of any non-hypoglycemic seizure within the last two years, or ongoing treatment with anticonvulsants
* History of hypoglycemic seizures (grand-mal) or coma in the last year
* History of pheochromocytoma: fractionated metanephrines will be tested in patients with history increasing the risk for a catecholamine secreting tumor: Episodic or treatment refractory (requiring 4 or more medications to achieve normotension) hypertension, Paroxysms of tachycardia, pallor, or headache, Personal or family history of MEN 2A, MEN 2B, neurofibromatosis, or von Hippel-Lindau disease
* History of adrenal disease or tumor
* Hypertension with systolic BP ≥160 mm Hg or diastolic BP ≥100 despite treatment
* Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year), or treatment with anti-psychotic medications that are known to affect glucose regulation.
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting
* Established history of allergy or severe reaction to adhesive or tape that must be used in the study
* Use of oral (e.g. thiazolidinediones, biguanides, sulfonylureas, glitinides, DPP-4 inhibitors, SGLT-2 inhibitors) anti-diabetic medications
* Hemoglobin < 12 g/dl
* Any factors that, in the opinion of the principal investigator would interfere with the safe completion of the study

iLet Infusion Set Sub-Study

* Unable to provide informed consent (e.g. impaired cognition or judgment)
* Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of their insulin pump, impaired memory, unable to speak and read English)
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception
* Hemoglobin < 11 g/dl
* Unable to establish IV access, or subject reports difficult IV access in the past
* History of allergy or severe reaction to adhesive or tape that must be used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Diabetes Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be published as online supplemental material to the main paper describing the results, as we have done for all of our previous bionic pancreas studies.

RESULTS

PARTICIPANT FLOW:
Groups:
- iPhone BP First, Then iLet BP (Lilly gLucagon); iLet BP First, Then iPhone BP (Lilly Glucagon): iPhone based bionic pancreas using insulin lispro and Lilly glucagon. These visits will be conducted separately from the infusion set sub-study visits.
  iPhone bionic pancreas: An experimental device composed of three parts: a continuous glucose monitor, control algorithms running on an iPhone, and drug delivery using Tandem insulin pumps
  Lilly glucagon: An aqueous formulation of human glucagon with limited stability that must be changed daily
  iLet Bionic Pancreas using using insulin lispro and Lilly glucagon. These visits will be conducted separately from the infusion set sub-study visits.
  iLet bionic pancreas: An experimental device that combines the functions of the iPhone-based bionic pancreas into one device.
- iLet Infusion Set First, Then Contact Detach: The infusion set sub-study will be testing just the experimental iLet infusion set in a crossover with the contact detach infusion set. These visits will be conducted separately from the iPhone and iLet bionic pancreas visits.
  iLet infusion set: The infusion set sub-study will be studying the experimental iLet infusion set in a cross-over with the Contact Detach infusion set. These visits will be conducted separately from the iPhone and iLet BP visits.
  Contact Detach infusion set: The infusion set sub-study will be studying the experimental iLet infusion set in a cross-over with the Contact Detach infusion set. These visits will be conducted separately from the iPhone and iLet BP visits.
- Contact Detach Infusion Set First, Then iLet Infusion Set: The infusion set sub-study will be testing just the experimental iLet infusion set in a crossover with the contact detach infusion set. These visits will be conducted separately from the iPhone and iLet bionic pancreas visits.
  Contact Detach infusion set: The infusion set sub-study will be studying the experimental iLet infusion set in a cross-over with the Contact Detach infusion set. These visits will be conducted separately from the iPhone and iLet BP visits.
  iLet infusion set: The infusion set sub-study will be studying the experimental iLet infusion set in a cross-over with the Contact Detach infusion set. These visits will be conducted separately from the iPhone and iLet BP visits.
Period: Overall Study
Arm/Group | iPhone BP First, Then iLet BP (Lilly gLucagon) | iLet BP First, Then iPhone BP (Lilly Glucagon) | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set First, Then Contact Detach | Contact Detach Infusion Set First, Then iLet Infusion Set
Started | 6 | 6 | 0 | 4 | 4
Completed | 6 | 3 | 0 | 3 | 1
Not Completed | 0 | 3 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: The study was terminated and the iLet BP arm with Xeris glucagon was never conducted.
Groups:
- iPhone Bionic Pancreas - Lilly Glucagon: iPhone based bionic pancreas using insulin lispro and Lilly glucagon. These visits will be conducted separately from the infusion set sub-study visits.
  iPhone bionic pancreas: An experimental device composed of three parts: a continuous glucose monitor, control algorithms running on an iPhone, and drug delivery using Tandem insulin pumps Lilly glucagon: An aqueous formulation of human glucagon with limited stability that must be changed dailyy
- Contact Detach First, Then iLet Infusion Set: The infusion set sub-study will be testing just the experimental iLet infusion set in a crossover with the contact detach infusion set. These visits will be conducted separately from the iPhone and iLet bionic pancreas visits.
  Contact Detach infusion set: The infusion set sub-study will be studying the experimental iLet infusion set in a cross-over with the Contact Detach infusion set. These visits will be conducted separately from the iPhone and iLet BP visits.
  iLet infusion set: The infusion set sub-study will be studying the experimental iLet infusion set in a cross-over with the Contact Detach infusion set. These visits will be conducted separately from the iPhone and iLet BP visits.
- Total: Total of all reporting groups
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set First, Then Contact Detach | Contact Detach First, Then iLet Infusion Set | Total
Number analyzed (Participants) | 6 | 6 | 0 | 4 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (22.3) | 32.6 (17.9) |  | 48.8 (14.7) | 44.7 (17.7) | 39.7 (17.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 |  | 3 | 2 | 14
  Male | 1 | 2 |  | 1 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 |  | 3 | 4 | 19
  Unknown or Not Reported | 0 | 0 |  | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0 | 0 | 0
  Asian | 0 | 0 |  | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0 | 0 | 0
  Black or African American | 0 | 0 |  | 0 | 0 | 0
  White | 6 | 6 |  | 4 | 4 | 20
  More than one race | 0 | 0 |  | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 |  | 4 | 4 | 20
Hemoglobin A1c [Mean (Standard Deviation); unit: percent] | 8.3 (0.7) | 7.6 (1.8) |  | 6.9 (1.2) | 8.1 (1.8) | 7.8 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Average Percent Dose Amounts Calculated by the Bionic Pancreas Control Algorithm That Are Successfully Delivered by the Pump (Aggregate of Both Insulin and Glucagon Doses)
Description: Average percent dose amounts calculated by the bionic pancreas control algorithm that are successfully delivered by the pump (aggregate of both insulin and glucagon doses) - primary outcome for iPhone-based BP using Lilly glucagon vs. iLet BP using Lilly glucagon
Time Frame: 8 hours
Population: This analysis only applies to the iPhone BP vs iLet BP using Lilly glucagon arms. The experimental arm with the iLet BP using Xeris glucagon was never conducted. This analysis does not apply to the infusion set sub study. Analysis includes 9 subjects that completed both the BP visits.
Measure: Mean (Standard Deviation); unit: percentage of doses delivered
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
percentage of doses delivered | 94.6 (9.2) | 95.0 (12.3) |  |  |

2. Primary Outcome: Average Percent Dose Amounts Calculated by the Bionic Pancreas Control Algorithm That Are Successfully Delivered by the Pump (Glucagon Doses).
Description: Average percent dose amounts calculated by the bionic pancreas control algorithm that are successfully delivered by the pump (glucagon doses) - - primary outcome for iLet BP using Lilly glucagon vs. iLet BP using Xeris Xerisol glucagon
Time Frame: 8 hours
Population: This analysis only applies to the iLet BP using Lilly glucagon vs the iLet BP using Xerisol glucagon arms. The experimental arm with the iLet BP using Xeris glucagon was never conducted. Data for this outcome is reported for the iPhone BP and iLet BP arms using Lilly glucagon. This analysis does not apply to the infusion set sub study.
Measure: Mean (Standard Deviation); unit: percentage of doses
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
percentage of doses | 96.6 (6.8) | 100.0 (0.5) |  |  |

3. Primary Outcome: Insulin Area Under the Curve in the 3.5 Hours Following the Insulin Bolus
Description: This applies only to the infusion set sub-study
Time Frame: 3.5 hours following insulin bolus
Population: This outcome only applies to the infusion set sub study, the other arms were not analyzed. The infusion set sub study was terminated and the insulin assays were not completed.
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Average Continuous Glucose Monitor (CGM) Glucose
Description: The average glucose according to continuous glucose monitor readings. This only applies to the iPhone vs. iLet BP experiments.
Time Frame: 8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
mg/dl | 179.2 (37.5) | 251.2 (80.0) |  |  |

5. Secondary Outcome: Percentage of Time in Each of the Following Ranges: < 50 mg/dl, < 60 mg/dl, <70 mg/dl, 70-120 mg/dl, 70-180 mg/dl, >180 mg/dl, >250 mg/dl
Description: Percentage of time subjects spent in each of these ranges based on continuous glucose monitor readings. This only applies to the iPhone vs iLet BP visits.
Time Frame: 8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
percentage of time
  CGM glucose < 60 | 0.0 (0.0) | 0.36 (1.07) |  |  |
  CGM glucose > 180 | 39.0 (24.5) | 67.5 (21.3) |  |  |

6. Secondary Outcome: Number of Subjects With Mean CGM Glucose < 154 mg/dl
Description: The number of subjects who achieved a mean CGM glucose < 154 mg/dl, which correlates to an estimated hemoglobin a1c of 7%, which is the ADA goal for therapy. This applies only to the iPhone vs iLet BP experiments
Time Frame: 8 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
Participants | 1 | 1 |  |  |

7. Secondary Outcome: Number of Severe Hypoglycemic Events (Subject Unable to Self-treat, Requiring the Assistance of Another Person)
Description: The number of severe hypoglycemic events subjects experience. This applies only to the iPhone vs iLet BP experiments.
Time Frame: 8 hours
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
events | 0 | 0 |  |  |

8. Secondary Outcome: Average Percent Insulin Dose Amounts Calculated by the Bionic Pancreas Control Algorithm That Are Successfully Delivered by the Pump.
Description: The average percentage of successfully delivered insulin doses. This applies only to the iPhone vs iLet BP experiments.
Time Frame: 8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of doses
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
percentage of doses | 94.0 (10.7) | 95.8 (13.3) |  |  |

9. Secondary Outcome: Average Percent Glucagon Dose Amounts Calculated by the Bionic Pancreas Control Algorithm That Are Successfully Delivered by the Pump.
Description: The average percentage of successfully delivered glucagon doses. This applies only to the iPhone vs iLet BP experiments.
Time Frame: 8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of doses
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
percentage of doses | 96.6 (6.8) | 100.0 (0.5) |  |  |

10. Secondary Outcome: Average Percent Insulin Dose Amounts Successfully Issued to the Pump by the Bionic Pancreas Control Algorithm That Are Successfully Delivered by the Pump.
Description: The average percentage of successfully issued insulin doses that are then delivered successfully by the pump. This applies only to the iPhone vs iLet BP experiments.
Time Frame: 8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of doses
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
percentage of doses | 98.5 (5.5) | 96.1 (13.1) |  |  |

11. Secondary Outcome: Average Percent Glucagon Dose Amounts Successfully Issued to the Pump by the Bionic Pancreas Control Algorithm That a Successfully Delivered by the Pump.
Description: The average percentage of successfully issued glucagon doses that are then delivered successfully by the pump. This applies only to the iPhone vs iLet BP experiments.
Time Frame: 8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of doses
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
percentage of doses | 96.6 (6.8) | 100.0 (0.5) |  |  |

12. Secondary Outcome: Average Percent of 5 Minute Steps During Which the Bionic Pancreas is Functioning Nominally in All Respects Based on Real-time CGM Data (New CGM Glucose Reading Captured, Dose Calculated, Dose Issued to Pumps
Description: The percentage of time (measured in 5 minute "steps") that the bionic pancreas is working, indicated by the presence of a CGM reading, a successful dose calculation and successful issuing of a dose. This applies only to the iPhone vs iLet BP experiments.
Time Frame: 8 hours
Population: This analysis only applies to the iPhone BP vs iLet BP using Lilly glucagon arms. The experimental arm with the iLet BP using Xeris glucagon was never conducted.
Measure: Mean (Standard Deviation); unit: percentage of 5 minute steps
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
percentage of 5 minute steps | 88.9 (0.073) | 75.1 (0.196) |  |  |

13. Secondary Outcome: Average Percent of 5 Minute Steps During Which the Bionic Pancreas is Functioning Nominally With or Without a New CGM Glucose Reading Captured (Dose Calculated, Dose Issued to Pumps).
Description: The percentage of time (measured in 5 minute "steps") that the bionic pancreas is working even without a CGM reading being present, indicated by a successful dose calculation and successful issuing of a dose. This applies only to the iPhone vs iLet BP experiments.
Time Frame: 8 hours
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage of 5 minutes steps
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
percentage of 5 minutes steps | 94.6 (0.054) | 99.8 (0.004) |  |  |

14. Secondary Outcome: CGM Reliability Index, Calculated as Percent of Possible Values Actually Recorded by CGM.
Description: A measure of CGM reliability, indicating the percentage of values the CGM displayed out of the total values it should have displayed in that time. This applies only to the iPhone vs iLet BP experiments.
Time Frame: 8 hours
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage of CGM values
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
percentage of CGM values | 94.1 (0.06) | 75.1 (0.19) |  |  |

15. Secondary Outcome: Glucagon Total Delivery Per kg of Body Mass.
Description: The average total glucagon delivered by the bionic pancreas. This applies only to the iPhone vs iLet BP experiments.
Time Frame: 8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
mcg/kg | 0.60 (0.84) | 1.12 (1.71) |  |  |

16. Secondary Outcome: Insulin Total Delivery Per kg of Body Mass.
Description: The average total insulin delivered by the bionic pancreas. This applies only to the iPhone vs iLet BP experiments.
Time Frame: 8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
units/kg | 0.22 (0.07) | 0.23 (0.07) |  |  |

17. Secondary Outcome: Number of Episodes of Symptomatic Hypoglycemia.
Description: Number of time subjects experienced symptoms of hypoglycemia and reported that to study staff. This applies only to the iPhone vs iLet BP experiments.
Time Frame: 8 hours
Population: as for outcome 1
Measure: Number; unit: number of episodes
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
number of episodes | 0 | 0 |  |  |

18. Secondary Outcome: Total Grams of Carbohydrate Taken for Hypoglycemia.
Description: The total grams of carbohydrates given to subjects for treatment of hypoglycemia. This applies only to the iPhone vs iLet BP experiments.
Time Frame: 8 hours
Population: as for outcome 1
Measure: Number; unit: number of grams of carbohydrates
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
number of grams of carbohydrates | 0 | 0 |  |  |

19. Secondary Outcome: Difference in Mean Nausea From VAS During the Study
Description: This applies only the iPhone vs. iLet BP experiments. Subjects were given a visual analog scale measuring 100 mm and asked to draw a line to indicate their level of nausea at timepoints during the study with 100 being the "worst possible nausea" and 0 being "no nausea".
Time Frame: 8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
score on a scale | 3.47 (10.47) | 6.93 (15.29) |  |  |

20. Secondary Outcome: Average Insulin Infusion Site Pain From VAS
Description: This applies to the iPhone vs. iLet BP experiments and the infusion set sub-study experiments. Subjects were given a visual analog scale measuring 100 mm and asked to draw a line to indicate their level of pain at timepoints during the study with 100 being the "worst possible pain" and 0 being "no pain".
Time Frame: 8 hours
Population: The experimental arm with the iLet BP using Xeris glucagon was never conducted. Analysis includes 9 subjects that completed both the BP visits and 4 subjects that completed both infusion set sub study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 4 | 4
score on a scale | 1.49 (3.06) | 6.61 (13.04) |  | 0.54 (2.61) | 2.42 (9.98)

21. Secondary Outcome: Difference in Local Erythema and Edema According to the Draize Scale
Description: This applies to the iPhone vs. iLet BP experiments and the infusion set sub-study experiments. The draize scale assess erythema, eschar and edema using a score from 0-4, with 4 meaning a worse outcome.
Time Frame: 8 hours
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 4 | 4
score on a scale | 0 (0) | 0 (0) |  | 0 (0) | 0 (0)

22. Secondary Outcome: Number of Unscheduled Infusion Set Replacements.
Description: This applies to the iPhone vs. iLet BP experiments and the infusion set sub-study experiments.
Time Frame: 8 hours
Population: as for outcome 20
Measure: Number; unit: number of infusion set changes
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 4 | 4
number of infusion set changes | 1 | 0 |  | 0 | 0

23. Secondary Outcome: Number of Unscheduled CGM Sensor Changes.
Description: This applies only to the iPhone vs. iLet BP experiments
Time Frame: 8 hours
Population: as for outcome 1
Measure: Number; unit: number of sensor changes
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0
number of sensor changes | 0 | 0 |  |  |

24. Secondary Outcome: Insulin Area Under the Curve During the Initial 90 Minute Fasted Period
Description: This applies only to the infusion set sub-study
Time Frame: 8 hours
Population: as for outcome 3
Arm/Group | iPhone BP First, Then iLet BP (Lilly gLucagon) | iLet BP First, Then iPhone BP (Lilly Glucagon) | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Mean Insulin Levels During the Initial 90 Minute Fasted Period
Description: This applies only to the infusion set sub-study
Time Frame: 8 hours
Population: as for outcome 3
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Difference Between Insulin Levels at Baseline and at 90 Minutes
Description: This applies only to the infusion set sub-study
Time Frame: 8 hours
Population: as for outcome 3
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Tmax After the Insulin Dose
Description: This applies only to the infusion set sub-study
Time Frame: 8 hours
Population: as for outcome 3
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: T 1/2 Max After the Insulin Dose
Description: This applies only to the infusion set sub-study
Time Frame: 8 hours
Population: as for outcome 3
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: C Max After the Insulin Dose
Description: This applies only to the infusion set sub-study
Time Frame: 8 hours
Population: as for outcome 3
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: AUC in the First 30 Minutes After the Insulin Dose
Description: This applies only to the infusion set sub-study
Time Frame: 8 hours
Population: as for outcome 3
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: AUC in the First 60 Minutes After the Insulin Dose
Description: This applies only to the infusion set sub-study
Time Frame: 8 hours
Population: as for outcome 3
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: AUC in the First 90 Minutes After the Insulin Dose
Description: This applies only to the infusion set sub-study
Time Frame: 8 hours
Population: This outcome only applies to the infusion set sub study, the other arms were not analyzed.The infusion set sub study was terminated and the insulin assays were not completed.
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

33. Secondary Outcome: Terminal Half Life After the Insulin Dose
Description: This applies only to the infusion set sub-study
Time Frame: 8 hours
Population: as for outcome 3
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

34. Secondary Outcome: Difference Between the Fasted PG Value and the PG Value at 90 Minutes
Description: This applies only to the infusion set sub-study
Time Frame: Baseline Fasted State and 90 Minutes
Population: This outcome only applies to the infusion set sub study, the other arms were not analyzed. The Overall Number of Participants Analyzed represents all Completed participants that received the intervention
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 4
mg/dl |  |  |  | -3.7 (28.7) | -6.7 (41.8)

35. Secondary Outcome: Difference in the PG Prior to the Meal and Peak Post-prandial Glucose
Description: This applies only to the infusion set sub-study
Time Frame: Pre-meal PG value and peak PG value during the 3.5 hours following the meal.
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 4
mg/dl |  |  |  | 176.3 (88.2) | 73.9 (76.8)

36. Secondary Outcome: PG AUC in the 3.5 Hours Following the Meal
Description: This applies only to the infusion set sub-study
Time Frame: 3.5 hours following the meal
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: mg*min/dl
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach Infusion Set
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 4
mg*min/dl |  |  |  | 15512740 (10050495) | 8359871 (5458714)

ADVERSE EVENTS:
Time Frame: During study visits up to 8 hours long
Description: There were no participants at risk for Serious Adverse Events, All-Cause Mortality and any other adverse events in the arm using the iLet bionic pancreas with Xerisol glucagon, because that arm was not conducted.
Groups:
- iPhone Bionic Pancreas - Lilly Glucagon: iPhone based bionic pancreas using insulin lispro and Lilly glucagon. These visits will be conducted separately from the infusion set sub-study visits.
  iPhone bionic pancreas: An experimental device composed of three parts: a continuous glucose monitor, control algorithms running on an iPhone, and drug delivery using Tandem insulin pumps Lilly glucagon: An aqueous formulation of human glucagon with limited stability that must be changed daily
- Contact Detach: Contact Detach infusion set: The infusion set sub-study will be studying the experimental iLet infusion set in a cross-over with the Contact Detach infusion set. These visits will be conducted separately from the iPhone and iLet BP visits.
Arm/Group | iPhone Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Lilly Glucagon | iLet Bionic Pancreas - Xerisol Glucagon | iLet Infusion Set | Contact Detach
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12 | 0/0 | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12 | 0/0 | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 7/12 | 0/0 | 0/5 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iPhone Bionic Pancreas - Lilly Glucagon (N=9) | iLet Bionic Pancreas - Lilly Glucagon (N=12) | iLet Bionic Pancreas - Xerisol Glucagon (N=0) | iLet Infusion Set (N=5) | Contact Detach (N=7)
Hyperglycemia (Endocrine disorders) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) — Hyperglycemia (may or may not include associated ketosis and vomiting) found to be associated with insulin infusion set failure

LIMITATIONS AND CAVEATS:
The original planned experiments and infusion set sub study were terminated early due to infusion site failures before the planned cohorts were completed. Changes to the infusion set design will be implemented prior to initiating any future studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT02701257/Prot_SAP_000.pdf